CLINICAL TRIAL: NCT06080633
Title: Research on Facial Prediction Technology for Edentulous Implant-Supported Fixed Prostheses Based on Multimodal Data Fusion
Brief Title: Facial Prediction Technology for Edentulous Patients
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Hongyang Ma, Research Associate, KU Leuven
Other Study IDs: S20230825
Record Dates: First submitted 2023-08-29; First posted 2023-10-12 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Edentulous Jaw
Keywords: Edentulous Jaw; deep learning; oral implantology; facial prediction
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to data from the World Health Organization, approximately 160 million people worldwide are edentulous. The incidence increases with age, and the proportion of edentulous patients is higher in the population aged 60 and above. Loss of teeth or edentulism can affect facial appearance, causing people to feel self-conscious and loss confidence in social situations, and even lead to psychological illnesses. Therefore, edentulous patients not only pay close attention to the recovery of oral function but also attach great importance to facial contour improvement. For a long time, due to technological limitations, clinicians have been unable to depict the changes in facial contour after implant placement for patients before surgery. However, with the development of artificial intelligence technology, deep learning-based methods for predicting soft tissue facial deformation have made this mission a possibility. This study established a multi-modal dataset for edentulous patients before and after implant restoration to lay the foundation for predicting facial contour changes after implant treatment. A graph generative adversarial network based on multi-modal data was proposed to achieve fast and high-precision facial contour prediction. To address the common challenges of slow computation and excessive computational resource consumption in current triangular mesh deformation simulation methods, this project innovatively proposed a graph generative adversarial network that uses multi-modal data and incorporates self-attention mechanisms to achieve fast and high-precision facial contour prediction for edentulous patients after implant restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete edentulism,
* aged 50 years or above,
* in good physical health,

Exclusion Criteria:

* patients who refuse to participate in the study，
* patients who cannot undergo facial scanning.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Edentulous Maxilla after Implant Prosthetic Restoration
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Soft Tissue Volume in the Lip Region after Implant Dentistry | Between pre-operation and after Implant-Supported Fixed Prostheses up to 3 months
  Quantitative analysis of lip volume changes in patients after oral implant surgery using facial scanning equipment

CONTACTS AND LOCATIONS:
Locations (1):
- Hongyang Ma, Leuven, Heverlee, Belgium